CLINICAL TRIAL: NCT05995106
Title: Prospective Validation of Usefulness in the Hypertensive Disorder of Pregnancy With Cardiovascular Disease Management Solution Based on Interconnection to Hospital Examination
Brief Title: mHealth for Hypertensive Disorder of Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jung-Won Suh, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-2308-844-302
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Hypertensive Disorder of Pregnancy; Preeclampsia
MeSH Terms: conditions — Toxemia; Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App Group (Experimental): Patients assigned to the app group receive assistance from the research team to install the Heart4U application and familiarize themselves with its usage.
  Interventions: Other: Heart4U
- Usual Care Group (No Intervention): The app (n=290) and usual care groups (n-290) continue to receive active treatment as previously administered (guideline-based prenatal care).

INTERVENTIONS:
Other: Heart4U — Mobile app.
  Arms: App Group

SUMMARY:
Objectives: We have developed a cardiovascular disease management application named Heart4U, with the capability of integrating with the Electronic Medical Records (EMR) system within the hospital.

The main goal of this study is to evaluate the clinical effectiveness of a treatment approach that entails self-management of risk factors through a mobile application among pregnant individuals diagnosed with hypertensive cardiovascular conditions.

Methods: Patients assigned to the app group receive assistance from the research team to install the Heart4U application and familiarize themselves with its usage. Both the app group and the usual care group continue to receive active treatment as previously administered (guideline-based prenatal care). Follow-up observations occur at each obstetric examination prior to delivery and are conducted again at the first month postpartum. The primary endpoint of observation pertains to the difference in systolic blood pressure between the enrollment and study completion time points.

DETAILED DESCRIPTION:
Inclusion Criteria:

* Diagnosis: 1 or 2

  1. Pregnant women diagnosed with hypertensive disorders of pregnancy at or beyond 12 weeks of gestation:

     * Chronic hypertension: Diagnosed with hypertension within 20 weeks of gestation (elevated office/clinic blood pressure ≥140/90 mm Hg) or currently on antihypertensive medication.
     * Gestational hypertension: Newly diagnosed with hypertension after 20 weeks of gestation (elevated office/clinic blood pressure ≥140/90 mm Hg) or currently on antihypertensive medication.
     * Preeclampsia: Newly diagnosed with hypertension after 20 weeks of gestation (elevated office/clinic blood pressure ≥140/90 mm Hg) or currently on antihypertensive medication, and presents with proteinuria (300 mg/24 hours or urine protein-to-creatinine ratio ≥0.3), thrombocytopenia (less than 100,000 platelets per microliter), abnormal renal function (creatinine exceeding 1.1 or doubling of baseline), elevated liver enzymes (twice normal levels), neurological symptoms (headache, visual disturbances, seizures, etc.), and/or pulmonary edema.
     * Superimposed preeclampsia: Diagnosed with hypertension within 20 weeks of gestation (elevated office/clinic blood pressure ≥140/90 mm Hg) or currently on antihypertensive medication, and experiences symptoms or signs related to superimposed preeclampsia.
  2. Pregnant women at elevated risk for hypertensive disorders of pregnancy:

     Multifetal gestation, obesity, uncontrolled gestational or pre-existing diabetes, history of hypertensive disorder of pregnancy leading to preterm birth, presence of borderline blood pressure readings during antepartum care (elevated office/clinic blood pressure ≥130/80 mm Hg) following a previous diagnosis of hypertension-related disorder in a prior pregnancy.
* Adult individuals aged 18 years and above who possess a smartphone and are capable of independently utilizing the application, among pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: 1 or 2

  1. Pregnant women diagnosed with hypertensive disorders of pregnancy at or beyond 12 weeks of gestation:

     * Chronic hypertension: Diagnosed with hypertension within 20 weeks of gestation (elevated office/clinic blood pressure ≥140/90 mm Hg) or currently on antihypertensive medication.
     * Gestational hypertension: Newly diagnosed with hypertension after 20 weeks of gestation (elevated office/clinic blood pressure ≥140/90 mm Hg) or currently on antihypertensive medication.
     * Preeclampsia: Newly diagnosed with hypertension after 20 weeks of gestation (elevated office/clinic blood pressure ≥140/90 mm Hg) or currently on antihypertensive medication, and presents with proteinuria (300 mg/24 hours or urine protein-to-creatinine ratio ≥0.3), thrombocytopenia (less than 100,000 platelets per microliter), abnormal renal function (creatinine exceeding 1.1 or doubling of baseline), elevated liver enzymes (twice normal levels), neurological symptoms (headache, visual disturbances, seizures, etc.), and/or pulmonary edema.
     * Superimposed preeclampsia: Diagnosed with hypertension within 20 weeks of gestation (elevated office/clinic blood pressure ≥140/90 mm Hg) or currently on antihypertensive medication and experiences symptoms or signs related to superimposed preeclampsia.
  2. Pregnant women at elevated risk for hypertensive disorders of pregnancy:

     Multifetal gestation, obesity, uncontrolled gestational or pre-existing diabetes, history of hypertensive disorder of pregnancy leading to preterm birth, presence of borderline blood pressure readings during antepartum care (elevated office/clinic blood pressure ≥130/80 mm Hg) following a previous diagnosis of hypertension-related disorder in a prior pregnancy.

     , and
* Adult individuals aged 18 years and above who possess a smartphone and are capable of independently utilizing the application among pregnant women.

Exclusion Criteria:

* Patients with evidence of delusions, confusion, or other cognitive disorders.
* Patients deemed difficult to conduct this study on by the researchers due to various reasons.
* Cases where device familiarity is significantly low, making data collection challenging.
* Pregnant patients requiring immediate electronic fetal monitoring or maternal monitoring due to imminent delivery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
delta SBP | between at the time of enrollment and one month postpartum
  Systolic Blood pressure (SBP) difference

SECONDARY OUTCOMES:
Blood pressure (systolic, diastolic, mean) trajectory | between at the time of enrollment and one month postpartum
  BP measured at each visit
obstetric outcomes | between at the time of enrollment and one month postpartum
  (The use of antihypertensive medication, progression to eclampsia or preeclampsia, pulmonary edema, fetal growth restriction, oligohydramnios, premature placental abruption, preterm birth (delivery between 20 and less than 37 weeks of gestation)
Body mass index (kg/m2) trajectory | between at the time of enrollment and one month postpartum
  BP measured at each visit
trajectory of the recorded step counts | between at the time of enrollment and one month postpartum
  on a pedometer application within a mobile phone.
Depression evaluation questionnaire | at the time of enrollment and one month postpartum
  Patient health questionnaires-9, Beck Depression Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Won Suh, MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Background] Kang SH, Baek H, Cho J, Kim S, Hwang H, Lee W, Park JJ, Yoon YE, Yoon CH, Cho YS, Youn TJ, Cho GY, Chae IH, Choi DJ, Yoo S, Suh JW. Management of cardiovascular disease using an mHealth tool: a randomized clinical trial. NPJ Digit Med. 2021 Dec 3;4(1):165. doi: 10.1038/s41746-021-00535-z. PMID 34862449
- [Derived] Kwun JS, Choi J, Yoon YE, Choi HM, Park JY, Kim HJ, Lee MJ, Choi BY, Yoo S, Suh JW. Prospective validation of a mobile health application for blood pressure management in patients with hypertensive disorders of pregnancy: study protocol for a randomized controlled trial. Trials. 2024 Jul 2;25(1):435. doi: 10.1186/s13063-024-08200-y. PMID 38956675